CLINICAL TRIAL: NCT06576206
Title: Effects of Bin Therapy on Finger Gnosia and Fine Motor Skills in Children With Down Syndrome
Brief Title: Effects of Bin Therapy on Finger Gnosia And Fine Motor Skill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0798
Record Dates: First submitted 2024-06-11; First posted 2024-08-28 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Down Syndrome
Keywords: down syndrome; bin therapy; freely box activties; finger gnosia
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: it will be randomized control trial in which non probability convenient sampling will be used. Two groups of age 6-12 will be formed in which participants will be randomly divided. Group A will receive conventional physical therapy exercise program including core strengthening, balance and coordination exercise, fine motor activities and group b will receive BIN therapy and finger gnosia
Who Masked: Participant
Masking Description: participants will get separate treatment protocols and possible efforts will be put to mask the the both group about treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physical therapy (Experimental): Control Group
  Interventions: Other: conventional therapy
- bin therapy and finger gnosia (Experimental): Experimental Group
  Interventions: Other: Bin therapy and finger gnosia

INTERVENTIONS:
Other: Bin therapy and finger gnosia — Schedule bin therapy sessions 2-3 times per week at first, increasing the frequency as participants get used to it. Data will be collected twice i.e., at the start of the study and after completion of 6 weeks of treatment by using outcome measure tools
  Arms: bin therapy and finger gnosia
Other: conventional therapy — schedule conventional therapy with 20-50 minutes of each session with each set comprises of 10-12 repetitions of each exercise
  Arms: conventional physical therapy

SUMMARY:
Down syndrome is a hereditary disorder resulting from the occurrence of an additional copy of chromosome 21, resulting in discernible variations in cognitive and physical characteristics. Finger gnosis pertains to the capacity to identify and discriminate among individual fingers. Tactile perception and body awareness are both encompassed by this particular component. Finger gnosis encompasses the sensory and cognitive mechanisms that enable an individual to recognize, label, and differentiate between their own fingers and those belonging to others. The therapeutic approach known as BIN Therapy is a non-invasive and pharmacologically unassisted intervention that use electrical stimulation as a means to enhance manual dexterity in individuals afflicted with neurological conditions

DETAILED DESCRIPTION:
It will be a randomized controlled trial. 30 patients fulfilling the inclusion and exclusion criteria will be recruited by non-probability convenience sampling and then randomly divided in two groups using lottery method. Group A will receive will receive conventional physical therapy exercise program including core strengthening, balance and coordination exercise, fine motor skills activities with 2-3 times a week, with 20-50 minutes of each session with each set comprises of 10-12 repetitions of each exercise. And the group B will receive BIN therapy and finger gnosia. Sensory assessment will be assess by Revised Nottingham sensory assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 5-13 years
* Children with Down syndrome who are able to follow simple instructions.
* Medically stable participants can participate in therapeutic procedures.
* Participants and their families should be able to attend Bin Therapy weekly.

Exclusion Criteria:

* Any other medical conditions or cognitive impairments that could affect their participation in the study.
* History of seizures.
* History of heart problems

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Finger Gnosia Assessed by Vernier Caliper | baseline and 8th week
  Finger gnosia assessed by vernier caliper by two-point discrimination test. 2-5 mm average score, 6-10 mm mild impairment, 11-15 moderate impairment, 16 mm or above severe impairment

SECONDARY OUTCOMES:
Nottingham sensory assessment | baseline and 8th weeks
  tactile sensation 42 max score, proprioception and Kinesthesia 24 max score, total score 66- 0-20 severe sensory impairment, 21-40 moderate sensory impairment, 41-54 mild sensory impairment, 55 - 66 normal sensory function

CONTACTS AND LOCATIONS:
Overall Officials: Hafsa Yasin, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischer U, Suggate SP, Stoeger H. Fine motor skills and finger gnosia contribute to preschool children's numerical competencies. Acta Psychol (Amst). 2022 Jun;226:103576. doi: 10.1016/j.actpsy.2022.103576. Epub 2022 Apr 4. PMID 35390583